CLINICAL TRIAL: NCT00970827
Title: Remote Ischemic Postconditioning During Percutaneous Coronary Interventions.
Acronym: RIP-PCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shahar Lavi, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R-09-015; 15664 (Other: REB)
Record Dates: First submitted 2009-07-09; First posted 2009-09-03 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; PCI; Postconditioning; Elective or urgent PCI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Leg postconditioning
  Interventions: Procedure: remote ischemic postconditioning
- 2 (Active Comparator): Arm postconditioning
  Interventions: Procedure: remote ischemic postconditioning
- 3 (Placebo Comparator): Control group
  Interventions: Procedure: remote ischemic postconditioning

INTERVENTIONS:
Procedure: remote ischemic postconditioning — Three 5- minute cycles of blood pressure cuff inflation according to the assigned group. The cuff is inflated to 200 mm Hg (and at least 20 mmHg above the systolic blood pressure) for 5 minutes followed by a 5-minute deflation (reperfusion).

SUMMARY:
Angioplasty is a commonly performed procedure for treating blockage of the blood vessels in the heart. Although this procedure is usually successful, it is often accompanied by a small degree of damage to the heart (i.e., small heart attack).

The purpose of this study is to find out if inflating a blood pressure cuff on the arm or the leg at the time of angioplasty for several minutes has a beneficial effect.

Patients will be assigned to one of three treatment groups: inflating blood pressure cuff on the arm, inflating blood pressure cuff on the leg and a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for PCI

Exclusion Criteria:

* Acute myocardial infarction
* Myocardial infarction or coronary bypass surgery during the last 4 weeks before PCI
* Use of Glyburide
* Heart failure (NYHA III/IV)
* Chronic inflammatory disease
* Severe renal impairment
* Significant peripheral vascular disease
* Unsuitable for use of an embolic protection device for PCI to SVG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2009-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Myocardial injury after PCI. | 24 hours

SECONDARY OUTCOMES:
To study the effects of different degrees of remote ischemic postconditioning on myocardial necrosis and inflammation following PCI. | 24 hours
Platelet function | 24 hours
Cardiac events | One year

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Lavi, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sceinces Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Lavi S, Abu-Romeh N, Wall S, Alemayehu M, Lavi R. Long-term outcome following remote ischemic postconditioning during percutaneous coronary interventions-the RIP-PCI trial long-term follow-up. Clin Cardiol. 2017 May;40(5):268-274. doi: 10.1002/clc.22668. Epub 2017 Jan 11. PMID 28075499
- [Derived] Lavi S, D'Alfonso S, Diamantouros P, Camuglia A, Garg P, Teefy P, Jablonsky G, Sridhar K, Lavi R. Remote ischemic postconditioning during percutaneous coronary interventions: remote ischemic postconditioning-percutaneous coronary intervention randomized trial. Circ Cardiovasc Interv. 2014 Apr;7(2):225-32. doi: 10.1161/CIRCINTERVENTIONS.113.000948. Epub 2014 Apr 1. PMID 24692535